CLINICAL TRIAL: NCT05632445
Title: Antithrombotic Therapy After Left Atrial Appendage Occlusion: Double Antiplatelet Therapy vs Apixaban
Brief Title: Apixaban vs Dual Antiplatet Therapy Study After Left Atrial Appendage Occlosure (ADALA)
Acronym: ADALA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DR. XAVIER FREIXA (Other)
Responsible Party: Sponsor-Investigator, DR. XAVIER FREIXA, MD; PhD. Interventional Cardiologist. Principal Investigator, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CV 185-685
Record Dates: First submitted 2022-08-05; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Left Atrial Appendage Occlusion
Keywords: Left atrial appendage occlusion, atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban (Other): Apixaban 5mg bid oral.Duration: 3 months Aspirin 80 / 100 mg bid oral. Duration: 9 months
  Interventions: Drug: Apixaban vs. DAPT
- DAPT (Other): Aspirin 80/100 mg + Clopidogrel 75 mg bid oral. Duration: 3 months Aspirin 80 / 100 mg bid oral. Durtaion: 9 months
  Interventions: Drug: Apixaban vs. DAPT

INTERVENTIONS:
Drug: Apixaban vs. DAPT — Apixaban vs DAPT after LAAO

SUMMARY:
Objective: To demonstrate superiority of a strategy of anticoagulation with apixaban 5mg/2.5mg bid as compared with the current standard of care (dual antiplatelet therapy) after occlusion of the left atrial appendage (LAAC) in patients with atrial fibrillation (AF).

Rationale: Data on antithrombotic therapy after LAAC are scarce and no randomized evaluation has been performed to demonstrate what is the best antithrombotic strategy. LAAO in patients without contraindication to chronic anticoagulants (PROTECT-AF regimen) is a 6-week period of anticoagulation with warfarin associated with aspirin, followed by once daily clopidogrel (75 mg) and aspirin (81-325 mg) until the 6 months visit, then aspirin alone is continued indefinitely, as tested in the pivotal trials. LAAO is also being used as an alternative to warfarin anticoagulation when patients have a contraindication or are unsuitable to warfarin. These patients usually receive a regimen of daily clopidogrel and aspirin (DAPT) for 3 months. Some may receive a shorter duration of DAPT or even only single antiplatelet therapy (SAPT) in case of excess bleeding risk. This antiplatelet regimen has never been compared with any anticoagulation regimen after LAAC. The Investigators propose to evaluate a unique antithrombotic strategy after LAAC for atrial fibrillation, whatever the indication of LAAC, including patients not suitable for long term warfarin anticoagulation. This strategy uses apixaban 5mg (with dose adjustment when necessary) which will be compared to the standard of care based on antiplatelet therapy and which may vary according to the risk profile of the patient. Apixaban, has demonstrated a mortality benefit associated with significant reductions in stroke, systemic embolism and major bleeding versus VKA. In addition, apixaban is the only NOAC which has demonstrated superiority over aspirin alone, in AF patients not suitable for chronic warfarin anticoagulation, to prevent cardio-embolic events with a safety profile similar to aspirin.The Investigators therefore formulate the hypothesis that apixaban is superior to standard of care (APT) to prevent cardiovascular events and bleeding complications after LAAO.

Population: Inclusion criteria: AF patients who have undergone a successful LAAO procedure. Exclusion criteria include any indication for triple antithrombotic treatment, mechanical heart valve, use of prasugrel or ticagrelor, serious renal failure defined as a creatinine clearance <15mL/min, contraindication to any form of anticoagulation or antiplatelet therapy. Randomization will occur always before hospital discharge as soon as the patient is stable or stabilized after the procedure.

Randomization: Apixaban vs. APT, both for 3 months. Groups: 1/Apixaban 5mg or 2.5mg bid (if dose adjustment needed). 2/ DAPT using low-dose ASA (75-100mg) and clopidogrel (75mg); or in patients with a history of intracranial hemorrhage (ICH) SAPT (aspirin or clopidogrel) will be used instead of DAPT from the time of randomization.

Follow-up: 12 months from randomization Primary endpoint: combined enpoint of death, MI, stroke, thromboembolic complications, major or significant bleeding at 3 months follow-up.

Sample size: In order to find a 16% difference in the event rates among the two treatment strategies, using a logrank test with a 5% two-sided significance level, we will need 76 patients in each group (152 in total). However, to compensate patient drop out, a total of 160 patients will be included in the study.

Recruitment : 24 months Centers: 3 centers in Spain.

DETAILED DESCRIPTION:
The non-valvular atrial fibrillation (NVAF) is the most common rhythm disturbance in our midst. Its incidence is correlated with age; therefore a significant increase is expected in the coming years due to the progressive aging of the population. Moreover, NVAF is responsible for up to 20% of all ischemic strokes and implies a worse prognosis compared with stroke due to other etiologies1 Oral anticoagulation is the standard therapy on patients with NVAF to reduce embolic events. The new anticoagulant drugs (NOAC) including the direct thrombin inhibitors (dabigatran2) and Xa inhibitors (apixaban3 and rivaroxaban4) have revealed a more stable and secure profile comparing to vitamin K antagonist. However, these new molecules still have an increased risk of bleeding (annual rate of major and minor bleeding of 2.15 -3.6% and 15-20% respectively) that might limit the use in a large amount of patients. Indeed about 40% of patients with indication for OAC not receive despite the introduction of NOAC5.

Percutaneous closure of the left atrial appendage (LAA) is recommended by the guidelines for patients with NVAF and contraindication for oral anticoagulation6,7 The aim of the intervention is: first reducing strokes caused by thrombus originated in the LAA)and second suppression of antithrombotic therapy avoiding the risk of bleeding associated with use of these drugs.

There are two devices that have been used for LAA closure worldwide: the WatchmanTM system (Boston Scientific, Boston, Massachusetts, USA) and AmplatzerTM Cardiac Plug (ACP) (St. Jude Medical, Minneapolis, Minnesota, USA). The currently available data comes mainly from the only two existing randomized trials to date (PROTECT AF8 and PREVAIL9). In these two RCT, patients treated with the Watchman device showed not to be inferior in terms of mortality and thromboembolic events compared to those patients treated with oral anticoagulation. In these trials, patients eligible to oral anticoagulation and percutaneous LAA occlusion (LAAO) were included, an uncommon situation in routine clinical practice. Moreover, even those randomized to LAA closure were treated with warfarin for at least six weeks, making it difficult to assess the benefit of appendage closure in early stages..

The ACP is a self-expanding device specifically designed to completely cover the ostium of the appendage. It comprises a nitinol lobe and a disk connected by a central waist. There are no randomized controlled trials with this device, but there is a large experience in registries including mainly patients with formal contraindication to OAC10,11 Despite the growing evidence about this technique, there are several questions that need to be answered: 1) Device thrombosis is a rare complication, but it has been described with the both devices (Watchman and ACP) 10-13. The incidence of device thrombosis is ranging between 2 and 17%, this wide variation might be due to misdiagnosis in some series since the incidence is higher in those series were more TEE were performed13,14. The relevance of device thrombosis is unclear; some series have showed a lack of correlation between the presence of device thrombosis and stroke (i0.3% of thrombosis have clinical translation) 12-14, but the experience its limited and device thrombosis and stroke remain as one of the most feared complications. 2) The presence of peri-device leaks during follow-up still has an uncertain meaning and makes difficult the decision of stopping antithrombotic therapy. In the surgical experience with appendage excision during mitral valve surgery, it was observed that incomplete excision of the OI was associated with a higher rate of embolic events. However, LAA percutaneous occlusion (LAAO) publications have not showed a clear relation between the presence of leaks and clinical events (stroke or device thrombosis)14,15. 3) Another point of controversy lies in the antithrombotic recommendations following the procedure. Since most of device thrombosis occur during the first trimester after closure and have been successfully treated with heparin or LWMH, the use of oral anticoagulation during the initial phase has been postulated 8,9. However, most of the patients treated with LAAO have a high risk of bleeding, and since the incidence and embolic potential of device thrombosis remains unclear, it makes difficult to justify the use of anticoagulation on this patients. In the other hand, dual antiplatelet therapy (DAT) has been used based on the prior experience with coronary stents. However, despite revealing a low device thrombosis and stroke rate, this protocol has not shown a reduction on major bleeding12,14-16.

In summary, the best antithrombotic therapy after LAA closure needs to provide a balance between efficacy (for prevention of thrombosis device) and safety (for the occurrence of major bleeding). Mainly because patients treated with therapy show a high risk for thromboembolic events (CHADS high) and concomitantly, a high incidence of haemorrhagic events (high HASBLED). According to data from large LAA closure registries14,16 the main indications for appendage closure are gastrointestinal and intracranial bleeding, therefore patients with absolute or relative contraindication for OAC. The rate of intracranial or gastrointestinal bleeding with DAT is up to 7%, being even higher than OAC 17,18. With the aim of reducing the risk of bleeding, LAA closure protocols have tried to reduce the DAT to 3 months, but with no solid evidence. Meanwhile, the introduction of NOAC has opened a new spectrum of therapeutic options. Among this new generation of antithrombotic molecules Apixaban has shown a really good safety and efficacy profile with low rate of ischemic and haemorrhagic events3. Moreover, Apixaban has already been use to treat LAA and device thrombosis with success19. In this regard, we believe that Apixaban would improve the rates of efficacy (reducing device thrombosis) and safety (with lower rate of bleeding) compared to DAT after LAA percutaneous closure. In fact, antithrombotic therapy post-LAAO is not given to treat any thrombus; it is given just to prevent its formation. In this sense, both 2.5 mg and 5 mg/12h of Apixaban have shown in terms of deep vein thrombosis (DVT) prevention20 and even the low dose of Apixaban has been shown effective to treat LAA thrombus21 . Since some patients undergoing LAAO present an extremely fragile profile and many patients have bled with different OAC strategies, including NOACs, we propose a strategy of 2.5 or 5 mg/12h of Apixaban based on the expected bleeding risk as this would provide the best balance between efficacy in preventing thrombus formation and avoid any kind of bleeding during the first 3 months after LAAO.

Hypothesis:

Treatment with Apixaban (5mg/12h or 2.5 mg/12h in specific cases) during the first 3 months followed by single antiplatelet aspirin 80-100 mg / day for 9 months after LAA closure will provide greater efficacy (for prevention of thromboembolic events clinical and device thrombosis) and safety (for the incidence of major bleeding) than treatment with dual antiplatelet therapy (aspirin + clopidogrel) during the first 3 months after followed by single antiplatelet aspirin 80-100 mg / day for 9 months. The rationale to implement a more intensive therapy during the first 3 months after LAAO responds to the period of higher risk of thrombus formation. Treatment duration (DAPT or apixaban for 3 months and then SAPT) is based on common clinical practice as described in the main LAAO registries (ACP multicenter registry, EWOLUTION or Amulet Observational study).

Objectives:

To demonstrate superiority of a strategy of anticoagulation with apixaban 5mg/2.5mg bid as compared with the current standard of care (dual antiplatelet therapy) after LAAO in patients with NVAF.

Primary end-point To compare the efficacy (for prevention of clinical thromboembolic events and device thrombosis) and safety (for the incidence of major bleeding) with Apixaban versus dual antiplatelet therapy (aspirin + clopidogrel) during the first 3 months after followed by single antiplatelet aspirin 80-100 mg / day for 9 months in both groups after LAA closure.

3- METHODS: The study will be conducted in accordance with good clinical practice and the institutional ethics committee in compliance with the protocol and with personnel who are qualified for every single duty.

Study design This is a phase IV multicenter randomized, open-label, controlled trial comparing the efficacy and safety of Apixaban vs. DAT after LAA occlusion (LAAO).

Inclusion Criteria:

* Age> 18 years
* NVAF (paroxysmal, persistent or permanent)
* CHADS2 score ≥1 or CHA2DS2-VASc score ≥2

  * Adequate anatomy for LAA closure and contraindication for OAC (absolute or relative).
* Able to give informed consent and to be followed-up (phone and clinical visit)

Exclusion criteria:

* Patients with mechanical prostheses, evidence of thrombus, complex aortic atheroma or symptomatic carotid disease
* Contraindication for TEE studies
* Platelets <40000
* Absolute contraindication to Apixaban for 3 months (severe renal failure with Cl. creat <15 ml / h or severe liver disease Child B or C) or allergy to the drug.

Contraindication to any form of anticoagulation or antiplatelet therapy.

* Patients with a history of drug or alcohol abuse, or psychosocial reasons that preclude the follow-up of the patient.
* Women of childbearing potential (WOCB) (See page .

End-Points:

Primary:

- Combined of efficacy (thromboembolic events prevention and device thrombosis) and safety (major bleeding incidence) at 3 months with both strategies.

Secondary:

* Combined of efficacy (thromboembolic events prevention and device thrombosis) and safety (major bleeding incidence) at 12 months with both strategies.
* Device thrombosis differences between the two strategies.
* Major bleeding differences between the two strategies.
* Any bleeding differences between the two strategies.

Study Protocol:

After establishing the indication for LAAO, a transesophageal echocardiography (TEE) will be performed in order to rule out intra-cardiac thrombus and measure/assess the LAA anatomy.

If the patient is a valid clinical and anatomical candidate for LAAO, the study will be explained and proposed and informed consent will be obtained. If the patient accepts and signs the consent, randomization will be performed after LAAO (see following sections). Baseline characteristics, general laboratory tests as well as basic physical examination will be performed and collected before randomization.

One hour before the intervention, prophylactic antibiotic will be administered (cephalosporin or vancomicin in case of betalactamic allergy). The procedure will be performed under general anesthesia or deep sedation and TEE guidance. Vascular access will be obtained from the right or left femoral vein and LAA access after transeptal puncture. Once left atrium access is achieved, a bolus of 100 IU/kg of ev heparin will be administered to reach an activated clotting tome (ACT) ≥250 seconds. If the patient was not under aspirin treatment before the intervention, a bolus of 1gr Inyesprin will be administered during the intervention. The procedure will be guided by fluoroscopy and TEE, which will allow additional LAA measuring, life time evaluation of catheters and device position as well as early detection of procedural complications such as pericardial effusion.

One day after the procedure a transthoracic echocardiography (TTE) will be performed in order to rule out pericardial effusion or device embolization. If there is no complication, patient will be discharged the following day.

Antithrombotic treatment:

Once LAAO is successfully performed, patient will be randomized 1:1 to one of the two treatment strategies. Randomization will be performed through a dedicated online website. For failed procedures (LAAO device not implanted), randomization will not be performed.

Four hours after the procedure and depending on the allocated treatment group patients will receive a first dose of apixaban (5 mg or 2.5mg*) or clopidogrel (600mg). Subsequently patients will receive:

Group 1: Apixaban* (5 or 2.5 mg/12h*) for the first 3 months after LAAO followed by aspirin 80-100 mg/day for 9 months.

Group 2: Aspirin 80-100 mg/day + clopidogrelª 75 mg/day followed by aspirin 80-100 mg/day for 9 months# *The standard dose of Apixaban will be 5 mg/12h unless the current product label does recommend use of lower apixaban dose (2.5 mg/12h). For the purpose of this study, use of 2.5mg/12h can be also considered in patients with expected increased bleeding risk (i.e. patients with previous bleeding with NOAC, patients with previous GI bleeding, patients with previous intracranial bleeding, patients with recurrent bleeding of any other territory) unless those patients fulfill absolute contraindications for use of apixaban. ** ª Patients with previous intracranial bleeding in Group 2 will receive aspirin 80-100 mg/day as single therapy.

It is understood that apixaban (5 and 2.5/12 h) will be provided and labelled by the company without additional costs. Storage, distribution and destruction process will be performed by the organizing centre.

At 12 months (out of the study), the treating physician will decide if he keeps aspirine indefinitely or stops it.

Follow-up:

Clinical follow-up will be performed at 1, 3, 6 and 12 months with a clinical visit and physical examination. The clinical visit will include specific assessment of thrombotic and bleeding events as well as general adverse events (AE) and serious adverse events (SAEs) (see appendix B) In these clinical visits we will specifically ask for concomitant treatments, discontinuation of subjects following any treatment with study drug, withdrawal of consent, drug overdose or risk of pregnancy.

At 3 and 12 months the Investigators will also collect general laboratory tests including hemoglobin, platelet count, coagulation status and renal function.

Imaging follow-up will include serial TEE or CT scan 1, 3 and 12 months after the index procedure in order to increase the sensitivity of device thrombosis detection. Since TEE/CT scan at 3 months is considered a standard of care after LAAO, only the 1 and 12 month TEE/CT scan could be considered additional diagnosis tests.

In case of any clinical thromboembolic event, device thrombosis or major bleeding (outcomes included in the primary outcome), antithrombotic treatment will be continued, stopped or changed according to the treating physician criteria.

Definitions:

The success of the procedure will be defined as implantation of the LAAO device without any major complication including death, stroke or any complication that requires surgical or endovascular treatment.

To evaluate procedural safety,the Investigators will include all clinical events within the hospitalization or the first 7 days after the procedure. For that purpose, clinical events will defined following the VARC consensus (Valve Academic Research Consortium)22 which includes: all- cause mortality, myocardial infarction, stroke (ischemic and hemorrhagic) or transient ischemic attack, systemic embolism, major bleeding and procedural complications such as device embolization, severe pericardial effusion or vascular complications. In addition, all other serious adverse events that occur following the subject´s written consent to participate in the study through 30 days of discontinuation of dosing will be reported to BMS Worlwide Safety The primary endpoint will only include events after hospitalization and at least 7 days after the index procedure in order to avoid the bias produced by potential complications during the procedure and not related to the medical treatment.

Major bleeding definition will be based on the Bleeding Academic Research Consortium23, corresponding to type 3 and 5: type 3a, bleeding with hemoglobin drop of 3 to 5 g/dl or need of blood transfusion; type 3b, bleeding with hemoglobin drop of >5 g/dl, cardiac tamponade, or bleeding requiring surgical intervention (skin, dental, nasal and hemorrhoid excluded) or intravenous vasoactive drugs; 3c, intracranial hemorrhage (micro-hematomas, intra-spinal or hemorrhagic transformation not included) or intraocular hemorrhage interfering with vision; type 5, mortal hemorrhage (type 5a, probable; type 5b, confirmed).

Device thrombosis will be defined as any thrombus with diameters >1mm and located over the LAAO device surface. Peri-device leaks will be classified according to the color jet width assessed by TEE 14: trivial (<1 mm), mild (1-3 mm), or relevant (> 3 mm). Complete LAAO will be defined as the absence of any relevant (>3mm) leak in the last TEE.

To evaluate the impact of the procedure in terms of stroke and bleeding prevention, the observed annual rate of events will be compared with the estimated rate based on the CHADS224, CHA2DS2-VASc24 and HAS-BLED25 scales.

Sample Size:

The sample size has been calculated based on the rate of observed events in the main LAAO registries with the ACP or Amulet devices. Considering the current indications for LAAC in Europe, our study population will be at much higher risk than the populations enrolled in the AF randomized studies (testing NOAC). In addition, the expected event rates are superior to the ones observed in the two main randomized studies (PROTECT AF and PREVAIL) as the target population has an absolute or relative contraindication to OAC. The Investigators have taken a rate for major or clinically significant bleeding of 15% in the DAPT group (control group) and an additional conservative rate of 10% for all ischemic end points, knowing that the Investigators consider also TIA, thrombosis on the device and PE events in our current composite endpoint (which were not accounted for in the cited studies. This makes a conservative 24% event rate per year for the primary endpoint over three months in the control group. Since the Investigators believe that apixaban will reduce both hemorrhagic and ischemic events, the Investigators expect an event rate between 8% and 10% in the apixaban group. In order to find a 16% difference in the event rates among the two treatment strategies, using a logrank test with a 5% two-sided significance level, the investigators will need 76 patients in each group (152 in total) with above 80% power. However, to compensate patient drop out, a total of 160 patients will be included in the study.

4- PROJECT VIABILITY: To include 160 patients, the investigators need to enroll three Spanish centers during a 2-year period. Each center should include a total of 53 patients (27 patients per year). Currently, there are several centers with that volume of LAAO and is expected to increase in the next years.

5- ADVERSE EVENT REPORTING All Serious Adverse Events (SAEs) that occur following the subject's written consent to participate in the study through 30 days of discontinuation of dosing must be reported to BMS Worldwide Safety.

Adverse Events:

An Adverse Event [AE] is defined as any new untoward medical occurrence or worsening of a pre existing medical condition in a patient or clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of investigational product, whether or not considered related to the investigational product.

The causal relationship to study drug is determined by a physician and should be used to assess all adverse events (AEs). The causal relationship can be one of the following:

Related: There is a reasonable causal relationship between study drug administration and the AE.

Not Related: There is not a reasonable causal relationship between study drug administration and the AE.

The term "reasonable causal relationship" means there is evidence to suggest a causal relationship.

Adverse events can be spontaneously reported or elicited during open-ended questioning, examination, or evaluation of a subject. (In order to prevent reporting bias, subjects should not be questioned regarding the specific occurrence of one or more adverse events).

Serious Adverse Events

A Serious Adverse Event (SAE) is any untoward medical occurrence at any dose that:

* results in death
* is life-threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
* requires inpatient hospitalization or causes prolongation of existing hospitalization (see NOTE*: below for exceptions)
* results in persistent or significant disability/incapacity
* is a congenital anomaly/birth defect
* is an important medical event, defined as a medical event that may not be immediately life-threatening or result in death or hospitalization but, based on appropriate medical and scientific judgment, may jeopardize the subject or may require intervention (e.g., medical, surgical) to prevent one of the other serious outcomes listed above. Examples of such events include but are not limited to intensive treatment in an emergency department or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization.
* Potential drug-induced liver injury (DILI) is also considered an important medical event--see the DILI section below for a definition of a potential DILI event.
* Suspected transmission of an infectious agent (eg, pathogenic or non-pathogenic) via the study drug is an SAE.
* Although pregnancy, overdose, and cancer are not always serious by regulatory definition, these events must be handled as SAEs.

  * NOTE: The following hospitalizations are not considered SAEs:

A visit to the emergency room or other hospital department lasting less than 24 hours that does not result in admission (unless considered an "important medical event" or a life-threatening event) Elective surgery planned before signing consent Admissions as per protocol for a planned medical/surgical procedure Routine health assessment requiring admission for baseline/trending of health status (eg, routine colonoscopy) Medical/surgical admission other than remedying ill health state that was planned before study entry. Appropriate documentation is required in these cases Admission encountered for another life circumstance that carries no bearing on health status and requires no medical/surgical intervention (eg, lack of housing, economic inadequacy, caregiver respite, family circumstances, administrative reason).

Adverse Events of Special Interest: In this study, the following adverse events are to be reported to BMS, regardless of wether these reports are classifed as serious or unexpected: Potential or suspected cases of liver injury including buit no limited to liver test abnormalities, jaundice, hepatitis or cholestasis

Adverse Events of Special Interest

In this study, the following adverse events are to be reported to BMS, regardless of whether these reports are classified as serious or unexpected:

Potential or suspected cases of liver injury including but not limited to liver test abnormalities, jaundice, hepatitis or cholestasis.

Serious Adverse Event Collecting and Reporting Following the subject's written consent to participate in the study, all SAEs, whether related or not related to study drug, must be collected, including those thought to be associated with protocol-specified procedures. All SAEs must be collected that occur during the screening period and within 30 days of discontinuing dosing. If applicable, SAEs must be collected that relate to any later protocol-specific procedure (such as follow-up skin biopsy).

The investigator should report any SAE occurring after these time periods that is believed to be related to study drug or protocol-specified procedure.

An SAE report should be completed for any event where doubt exists regarding its status of seriousness.

If the investigator believes that an SAE is not related to study drug, but is potentially related to the conditions of the study (such as withdrawal of previous therapy, or a complication of a study procedure), the relationship should be specified in the narrative section of the SAE Report Form.

SAEs, whether related or unrelated to the study drug, and pregnancies must be reported to BMS within 24 hours/1 business day after becoming aware of the event.. SAEs must be recorded on etiher CIOMS or approved site SAE form; Pregnancies must be reported and submitted to BMS on any of the following form(s): 1. CIOMS or 2. BMS Pregnancy Surveillance Form or, 3. Approved site SAE form.

SAE Email Address: Worldwide.Safety@BMS.com SAE Fax Number: 609-818-3804

If only limited information is initially available, follow-up reports are required. (Note: Follow-up SAE reports should include the same investigator term(s) initially reported.) If an ongoing SAE changes in its intensity or relationship to study drug or if new information becomes available, a follow-up SAE report should be sent within 24 hours to the BMS (or designee) using the same procedure used for transmitting the initial SAE report.

All SAEs should be followed to resolution or stabilization.

SAE Reconciliation The investigator will reconcile the clinical database SAE cases transmitted to BMS Global Pharmacovigilance (GPV&E). Frequency of reconciliation will be determined prior to study commencement but will occur no less than once prior to study database lock. BMS GPV&E will e-mail upon request from the investigator, the GPV&E reconciliation report. Requests for reconciliation should be sent to aepbusinessprocess@bms.com. The data elements listed on the GPV&E reconciliation report will be used for case identification purposes. If the investigator determines a case was not transmitted to BMS GPV&E, the case will be sent immediately.

All SAEs should simultaneously be faxed or e-mailed to BMS at:

Global Pharmacovigilance & Epidemiology Bristol-Myers Squibb Company Fax Number: 609-818-3804 Email: Worldwide.safety@bms.com

6- WOMEN OF CHILD-BEARING POTENTIAL (WOCBP)

Eligibility criteria must address WOCBP and their partners.

1. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
2. Women must not be breastfeeding
3. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) YY plus 5 half-lives of study drug YY (XX days) plus 30 days (duration of ovulatory cycle) for a total of XX days post-treatment completion.
4. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) YY plus 5 half-lives of the study drug (XX days) plus 90 days (duration of sperm turnover) for a total of XX days post-treatment completion.
5. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However they must still undergo pregnancy testing as described in this section.

Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

At a minimum, subjects must agree to the use of one method of highly effective contraception as listed below:

HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

* Male condoms with spermicide.
* Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena by WOCBP subject or male subject's WOCBP partnerFemale partners of male subjects participating in the study may use hormone based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug
* IUDs, such as ParaGard
* Tubal ligation
* Vasectomy.
* Complete Abstinence*

  * Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence

WOMEN OF CHILD-BEARING POTENTIAL (WOCBP) A Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40mIU/mL to confirm menopause.

* Females treated with hormone replacement therapy, (HRT) are likely to have artificially suppressed FSH levels and may require a washout period in order to obtain a physiologic FSH level. The duration of the washout period is a function of the type of HRT used. The duration of the washout period below are suggested guidelines and the investigators should use their judgement in checking serum FSH levels. If the serum FSH level is >40 mIU/ml at any time during the washout period, the woman can be considered postmenopausal :

  * 1 week minimum for vaginal hormonal products (rings, creams, gels)
  * 4 week minimum for transdermal products
  * 8 week minimum for oral products Other parenteral products may require washout periods as long as 6 months. Not Applicable.

    7- REQUESTED FUND (Purpose):

    1- Funding for study insurance. 2- Funding for financial support to centers for the work derived from the inclusion of patients and follow-up (additional clinical visits and TEE).

    3- Funding for centralized assessment (core-lab) of TEE during follow-up.

    8- STUDY BENEFITS

The Investigators strongly believe that a positive result in favor of apixaban would have a large impact on the scientific community as it would demonstrate the superiority of the drug compared to dual antiplatelet therapy in terms of efficacy and safety in a population with a high risk of both cardio-embolic and hemorrhagic events. In addition, apixaban would be used in a very specific setting like LAAO in which none of the other NOAC has been used.

It is very important to highlight that the present study does not try to show the superiority of LAAO over NOACS. In fact, it is the contrary as it might demonstrate that apixaban is very well tolerated in a population that has been categorized as not eligible for OAC.

ELIGIBILITY:
Inclusion Criteria:

* NVAF (paroxysmal, persistent or permanent)
* CHADS2 score >1 or CHA2DS2-VASc score >2
* Adequate anatomy for LAA closure and contraindication for OAC (absolute or relative).
* Able to give informed consent and to be followed -up (phone and clinical visit)

Exclusion Criteria:

* Patients with mechanical prostheses, evidence of thrombus, complex aortic atheroma or symptomatic carotid disease.
* Contraindication for TEE studies
* Platelets <40000
* Absolute contraindication to Apixaban for 3 months (severee renal failure with CI creat <15 ml/h or severe liver disease Child B or C) or allergy to the drug.
* Contraindication to any form of anticoagulation or antiplatelet therapy.
* Patients with a history of drug or alchol abuse, or psychosocial reasons that preclude the follow-up of the patient
* Women of childbearing potential (WOCB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Combined Safety-Efficacy at 3 months Apixaban vs dual antiplatelet therapy | 3 months
  Combined of efficacy (thromboembolic events prevention and device thrombosis) and safety (major bleeding incidence) at 3 months with both strategies.

SECONDARY OUTCOMES:
Combined Safety-Efficacy at 12 months apixaban vs dual antiplatelet therapy | 12 months
  Combined of efficacy (thromboembolic events prevention and device thrombosis) and safety (major bleeding incidence) at 12 months with both strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Dabit Arzamendi, Md, PhD, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Background] Connolly SJ, Eikelboom J, Joyner C, Diener HC, Hart R, Golitsyn S, Flaker G, Avezum A, Hohnloser SH, Diaz R, Talajic M, Zhu J, Pais P, Budaj A, Parkhomenko A, Jansky P, Commerford P, Tan RS, Sim KH, Lewis BS, Van Mieghem W, Lip GY, Kim JH, Lanas-Zanetti F, Gonzalez-Hermosillo A, Dans AL, Munawar M, O'Donnell M, Lawrence J, Lewis G, Afzal R, Yusuf S; AVERROES Steering Committee and Investigators. Apixaban in patients with atrial fibrillation. N Engl J Med. 2011 Mar 3;364(9):806-17. doi: 10.1056/NEJMoa1007432. Epub 2011 Feb 10. PMID 21309657
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Kirley K, Qato DM, Kornfield R, Stafford RS, Alexander GC. National trends in oral anticoagulant use in the United States, 2007 to 2011. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):615-21. doi: 10.1161/CIRCOUTCOMES.112.967299. Epub 2012 Sep 4. PMID 22949490
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines-CPG; Document Reviewers. 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation--developed with the special contribution of the European Heart Rhythm Association. Europace. 2012 Oct;14(10):1385-413. doi: 10.1093/europace/eus305. Epub 2012 Aug 24. No abstract available. PMID 22923145
- [Background] Meier B, Blaauw Y, Khattab AA, Lewalter T, Sievert H, Tondo C, Glikson M; Document Reviewers. EHRA/EAPCI expert consensus statement on catheter-based left atrial appendage occlusion. Europace. 2014 Oct;16(10):1397-416. doi: 10.1093/europace/euu174. Epub 2014 Aug 29. No abstract available. PMID 25172844
- [Background] Holmes DR, Reddy VY, Turi ZG, Doshi SK, Sievert H, Buchbinder M, Mullin CM, Sick P; PROTECT AF Investigators. Percutaneous closure of the left atrial appendage versus warfarin therapy for prevention of stroke in patients with atrial fibrillation: a randomised non-inferiority trial. Lancet. 2009 Aug 15;374(9689):534-42. doi: 10.1016/S0140-6736(09)61343-X. PMID 19683639
- [Background] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Background] Lam YY, Yip GW, Yu CM, Chan WW, Cheng BC, Yan BP, Clugston R, Yong G, Gattorna T, Paul V. Left atrial appendage closure with AMPLATZER cardiac plug for stroke prevention in atrial fibrillation: initial Asia-Pacific experience. Catheter Cardiovasc Interv. 2012 Apr 1;79(5):794-800. doi: 10.1002/ccd.23136. Epub 2011 Nov 30. PMID 21542102
- [Background] Reddy VY, Mobius-Winkler S, Miller MA, Neuzil P, Schuler G, Wiebe J, Sick P, Sievert H. Left atrial appendage closure with the Watchman device in patients with a contraindication for oral anticoagulation: the ASAP study (ASA Plavix Feasibility Study With Watchman Left Atrial Appendage Closure Technology). J Am Coll Cardiol. 2013 Jun 25;61(25):2551-6. doi: 10.1016/j.jacc.2013.03.035. Epub 2013 Apr 10. PMID 23583249
- [Background] Park JW, Bethencourt A, Sievert H, Santoro G, Meier B, Walsh K, Lopez-Minguez JR, Meerkin D, Valdes M, Ormerod O, Leithauser B. Left atrial appendage closure with Amplatzer cardiac plug in atrial fibrillation: initial European experience. Catheter Cardiovasc Interv. 2011 Apr 1;77(5):700-6. doi: 10.1002/ccd.22764. Epub 2011 Mar 8. PMID 20824765
- [Background] Lopez-Minguez JR, Eldoayen-Gragera J, Gonzalez-Fernandez R, Fernandez-Vegas C, Fuentes-Canamero ME, Millan-Nunez V, Nogales-Asensio JM, Martinez-Naharro A, Sanchez-Giralt S, Doblado-Calatrava M, Merchan-Herrera A. Immediate and one-year results in 35 consecutive patients after closure of left atrial appendage with the Amplatzer cardiac plug. Rev Esp Cardiol (Engl Ed). 2013 Feb;66(2):90-7. doi: 10.1016/j.rec.2012.04.017. Epub 2012 Aug 29. PMID 24775381
- [Background] Tzikas A, Shakir S, Gafoor S, Omran H, Berti S, Santoro G, Kefer J, Landmesser U, Nielsen-Kudsk JE, Cruz-Gonzalez I, Sievert H, Tichelbacker T, Kanagaratnam P, Nietlispach F, Aminian A, Kasch F, Freixa X, Danna P, Rezzaghi M, Vermeersch P, Stock F, Stolcova M, Costa M, Ibrahim R, Schillinger W, Meier B, Park JW. Left atrial appendage occlusion for stroke prevention in atrial fibrillation: multicentre experience with the AMPLATZER Cardiac Plug. EuroIntervention. 2016 Feb;11(10):1170-9. doi: 10.4244/EIJY15M01_06. PMID 25604089
- [Background] Freixa X, Tzikas A, Sobrino A, Chan J, Basmadjian AJ, Ibrahim R. Left atrial appendage closure with the Amplatzer Cardiac Plug: impact of shape and device sizing on follow-up leaks. Int J Cardiol. 2013 Sep 30;168(2):1023-7. doi: 10.1016/j.ijcard.2012.10.031. Epub 2012 Dec 27. PMID 23273340
- [Background] Urena M, Rodes-Cabau J, Freixa X, Saw J, Webb JG, Freeman M, Horlick E, Osten M, Chan A, Marquis JF, Champagne J, Ibrahim R. Percutaneous left atrial appendage closure with the AMPLATZER cardiac plug device in patients with nonvalvular atrial fibrillation and contraindications to anticoagulation therapy. J Am Coll Cardiol. 2013 Jul 9;62(2):96-102. doi: 10.1016/j.jacc.2013.02.089. Epub 2013 May 9. PMID 23665098
- [Background] Vidal-Jordana A, Barroeta-Espar I, Sainz Pelayo MP, Mateo J, Delgado-Mederos R, Marti-Fabregas J. [Intracerebral hemorrhage in anticoagulated patients: what do we do afterwards?]. Neurologia. 2012 Apr;27(3):136-42. doi: 10.1016/j.nrl.2011.04.020. Epub 2011 Jun 16. Spanish. PMID 21683480
- [Background] Healey JS, Hart RG, Pogue J, Pfeffer MA, Hohnloser SH, De Caterina R, Flaker G, Yusuf S, Connolly SJ. Risks and benefits of oral anticoagulation compared with clopidogrel plus aspirin in patients with atrial fibrillation according to stroke risk: the atrial fibrillation clopidogrel trial with irbesartan for prevention of vascular events (ACTIVE-W). Stroke. 2008 May;39(5):1482-6. doi: 10.1161/STROKEAHA.107.500199. Epub 2008 Mar 6. PMID 18323500
- [Background] Kawakami T, Kobayakawa H, Ohno H, Tanaka N, Ishihara H. Resolution of left atrial appendage thrombus with apixaban. Thromb J. 2013 Dec 20;11(1):26. doi: 10.1186/1477-9560-11-26. PMID 24359320
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. J Am Coll Cardiol. 2012 Oct 9;60(15):1438-54. doi: 10.1016/j.jacc.2012.09.001. PMID 23036636
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Lip GY, Frison L, Halperin JL, Lane DA. Identifying patients at high risk for stroke despite anticoagulation: a comparison of contemporary stroke risk stratification schemes in an anticoagulated atrial fibrillation cohort. Stroke. 2010 Dec;41(12):2731-8. doi: 10.1161/STROKEAHA.110.590257. Epub 2010 Oct 21. PMID 20966417
- [Background] Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010 Nov;138(5):1093-100. doi: 10.1378/chest.10-0134. Epub 2010 Mar 18. PMID 20299623
- [Result] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Derived] Freixa X, Cruz-Gonzalez I, Cepas-Guillen P, Millan X, Antunez-Muinos P, Flores-Umanzor E, Asmarats L, Regueiro A, Lopez-Tejero S, Li CP, Sanchis L, Rodes-Cabau J, Arzamendi D. Low-Dose Direct Oral Anticoagulation vs Dual Antiplatelet Therapy After Left Atrial Appendage Occlusion: The ADALA Randomized Clinical Trial. JAMA Cardiol. 2024 Oct 1;9(10):922-926. doi: 10.1001/jamacardio.2024.2335. PMID 39110427